CLINICAL TRIAL: NCT06229496
Title: A Phase 1b, Open-label, Multicenter, Dose Escalation and Dose Expansion Study of S-1 in Combination With Nab-paclitaxel and Gemcitabine (GAS) in Subjects With Metastatic Pancreatic Adenocarcinoma
Brief Title: Dose Escalation and Dose Expansion Study of GAS in Subjects With Metastatic Pancreatic Adenocarcinoma
Acronym: GAS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yeh Chun-Nan, Professor, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202300649A3
Record Dates: First submitted 2024-01-09; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: Dose escalation; Pancreatic adenocarcinoma; GAS
MeSH Terms: interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- GAS regimen-dose level 1 (Experimental)
  Interventions: Combination Product: Gemcitabine 800mg/m2 + Nab-paclitaxel 100mg/m2 + S-1 (dose according to BSA)
- GAS regimen-dose level 2 (Experimental)
  Interventions: Combination Product: Gemcitabine 800mg/m2 + Nab-paclitaxel 125mg/m2 + S-1 (dose according to BSA)
- GAS regimen-dose level 3 (Experimental)
  Interventions: Combination Product: Gemcitabine 1000mg/m2 + Nab-paclitaxel 125mg/m2 + S-1 (dose according to BSA)

INTERVENTIONS:
Combination Product: Gemcitabine 800mg/m2 + Nab-paclitaxel 100mg/m2 + S-1 (dose according to BSA) — Dose escalation study-dose level 1
  Arms: GAS regimen-dose level 1
Combination Product: Gemcitabine 800mg/m2 + Nab-paclitaxel 125mg/m2 + S-1 (dose according to BSA) — Dose escalation study-dose level 2
  Arms: GAS regimen-dose level 2
Combination Product: Gemcitabine 1000mg/m2 + Nab-paclitaxel 125mg/m2 + S-1 (dose according to BSA) — Dose escalation study-dose level 3
  Arms: GAS regimen-dose level 3

SUMMARY:
A Phase 1b, open-label, multicenter, dose escalation and dose expansion study of S-1 in combination with nab-paclitaxel and gemcitabine (GAS) in subjects with metastatic pancreatic adenocarcinoma. This study is a dose escalation and dose expansion study with the objective to establish the MTD and/or RP2D and/or DLT of nab-paclitaxel and gemcitabine in combination with a body surface area(BSA)-based dose of S-1 in subject with metastatic pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) is the seventh leading cause of cancer- related death worldwide as the second leading cause of cancer mortality in the United States by 2030 . The overall 5-year survival rate is around 5% for advanced PDAC and 15-30% for resected PDAC. While recent advances have emerged in precision medicine and immunotherapy in a variety of cancer types, unfortunately these drugs are not applicable to most patients with PDAC. To date, polychemotherapy combinations remain the mainstay of systemic treatments for advanced PDAC. Of note, FOLFIRINOX is a triplet combination regimen while nab-Paclitaxel and gemcitabine is a doublet combination. Both NALIRIFOX and FOLFIRINOX showed the same median OS with about 11.1 months from NAPOLI 3 and PRODIGE4 trials, respectively, demonstrating the biologically comparable anti-tumor effects. On the other hand, the median OS of 8.5 months of gemcitabine plus nab-paclitaxel raised the question-would it be possible to add the third active drug in this doublet combination to achieve more potential efficacy, being comparable with triplet combination such as FOLFIRINOX or NALIRIFOX. Therefore, in this study the investigator aimed to investigate whether adding S-1 to nab-paclitaxel and gemcitabine as GAS regimen can be a potential triplet combination.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed pancreatic adenocarcinoma (poorly differentiated carcinoma is allowed in the absence of neuroendocrine features or squamous differentiation)
2. Treatment-naï ve stage IV disease (measurable disease is required). Prior adjuvant chemotherapy or radiochemotherapy is allowed, if completed ≥ 6 months before enrollment.
3. Measurable disease defined as at least one lesion that can be measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan or MRI
4. Eastern Cooperative Oncology Group (ECOG) performance score of 0-1
5. Life expectancy > 6 months in the opinion of his/her treating physician.
6. At least 18 years of age
7. Ability to understand the nature of this study protocol, comply with study and/or follow-up procedures, and sign the IRB-approved written informed consent
8. Fertile female and male patients with child-bearing potential agree to use adequate contraceptive measures prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
9. Adequate bone marrow function:

   Absolute neutrophil count (ANC) ≥ 1500/uL Platelet count ≥ 100,000/uL Hemoglobin ≥ 9.0 g/dL
10. Adequate hepatic function:

    Total bilirubin ≤ 1.5 X ULN (≤3.5 mg/dL if with adequate biliary tract drainage/stent placement) AST ≤ 3.0 X ULN (≤5.0X ULN if liver metastases are present) ALT ≤ 3.0 X ULN (≤5.0X ULN if liver metastases are present)
11. Adequate renal function (defined as serum creatinine ≤ 1.5 X ULN or creatinine clearance rate (CCr) ≥ 50 mL/min (calculated by Cockroft-Gault formula; male: [(140 - age in years) × weight in kg)]/[72 × serum creatinine(mg/dL)];female=male x 0.85 )
12. Able to take the oral study medication (S-1)
13. No clinically significant abnormal ECG findings within 28 days (4 weeks) prior to enrollment

Exclusion Criteria:

1. Have known endocrine pancreatic tumors or ampullary cancer
2. Have received first line treatment for metastatic pancreatic cancer
3. Have a serious concomitant active infection or other major comorbidities that, in the opinion of the investigator, would compromise the patient's ability to adhere to the protocol (e.g., stroke, uncontrolled arrhythmia, heart failure, or active autoimmune disease)
4. Have HIV history or hepatitis B and C infection, except for prescribing anti-hepatitis B medications for hepatitis B carrier and undetectable HCV RNA level for hepatitis C prior to enrollment.
5. Have known central nervous system (CNS) malignancy or metastasis (screening is not required)
6. Have concurrent hematologic malignancies, acute or chronic leukemia
7. Have known additional malignancy that is progressing or required active treatments within the past 6 months, except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast or cervical cancer)
8. Women with a positive pregnancy test or who are breastfeeding
9. Have participated within the last 30 days in a clinical trial involving an investigational product
10. Unable to swallow capsules or has diseases significantly affecting gastrointestinal function or resection of the stomach or small bowel, malabsorption syndrome, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
11. Current peripheral sensory neuropathy ≥ Grade 2
12. Any social condition or diseases judged ineligible by physician for participation in the study due to safety concern

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | From cycle 1 day 1 (each cycle is 14 days) untill the date of radiographic tumor assessment confirm tumor recurrence or specified AE occur, assessed up to 3 years
  To determine a recommended Phase 2 dose (RP2D) of nab-paclitaxel and gemcitabine in combination with body surface area (BSA) - based dose of S-1 in subject with metastatic pancreatic adenocarcinoma
Dose-limiting toxicity (DLT) | From cycle 1 day 1 (each cycle is 14 days) untill the date of radiographic tumor assessment confirm tumor recurrence or specified AE occur, assessed up to 3 years
Objective response rate (ORR) | From cycle 1 day 1 (each cycle is 14 days) untill the date of radiographic tumor assessment confirm tumor recurrence or specified AE occur, assessed up to 3 years
  Tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1.

SECONDARY OUTCOMES:
Safety profile of GAS regimen | From cycle 1 day 1 (each cycle is 14 days) untill the date of radiographic tumor assessment confirm tumor recurrence or specified AE occur, assessed up to 3 years
  Safety profile will be recorded and graded according to NCI-CTCAE v 5.0.
Disease Control Rate (DCR) | Through study completion, an average of 3 year
  Defined as having complete response, partial response or stable disease at 12 weeks. (based on RECIST Version 1.1)
Duration of Response (DoR) | Through study completion, an average of 3 year
  Time from documentation of tumor response to disease progression. (based on RECIST Version 1.1)
Progression-free Survival (PFS) | Through study completion, an average of 3 year
  From the start date of study treatment to the date of progression disease or death. (based on RECIST Version 1.1)
Overall Survival (OS) | Through study completion, an average of 3 year
  From the start date of study treatment to the date of death.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Chang-Gung Memorial Hospital, Kaohsiung Branch, Kaohsiung City
  - Chang-Gung Memorial Hospital, Linkou Branch, Taoyuan District